CLINICAL TRIAL: NCT06713837
Title: IMPACT-AML: A Randomized Pragmatic Clinical Trial for Relapsed or Refractory Acute Myeloid Leukemia. IMPACT-AML RPCT
Brief Title: IMPACT-AML: A Randomized Pragmatic Clinical Trial for Relapsed or Refractory Acute Myeloid Leukemia.
Acronym: IMPACT-AML
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Collaborators: Hospital Vall d'Hebron (Other); Cyprus Institute of Neurology and Genetics (Other); European Leukemia Net (Unknown); Fundacion Para La Investigacion Hospital La Fe (Other); Ostdeutsche Studiengruppe Haematologie Und Onkologie e.V. (Unknown); Ospedale Pediatrico Bambin Gesù (Other); Czech Lymphoma Study Group (Other); Charite University, Berlin, Germany (Other); Fundación Instituto de Estudios de Ciencias de la Salud de Castilla y León (Other); University of Bologna (Other); Hannover Medical School (Other); German Society for Pediatric Oncology and Hematology GPOH gGmbH (Other); Toscana Life Sciences Sviluppo s.r.l. (Industry); Lithuanian University of Health Sciences (Other); Gruppo Italiano Malattie EMatologiche dell'Adulto (Other); TIMELEX (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRST204.07; 2024-514517-35-00 (EU CTIS Number); 101104421 (Other Grant/Funding Number: European Commission)
Record Dates: First submitted 2024-11-27; First posted 2024-12-03 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Acute Myeloid Leukemia; Relapse/Recurrence
Keywords: Relapsed/Refractory; Acute Myeloid Leukemia; Low Intensity therapy; Pragmatic; Low intervention Clinical trial; Randomized controlled trial; Horizon Europe; Mission Cancer; Diagnosis and treatment
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low intensity treatment (Experimental): Low intensity treatments are based on the single agent use of innovative and target drugs or their combination with other target drugs and less-toxic agents in doublets or triplets.
  Administration of low intensity therapies in combination with antibodies or target agents would be included in this cohort
  Interventions: Drug: Low intensity therapies
- High intensity treatment (Active Comparator): Intensive treatment of leukemia is based on high dose of chemotherapy agents.
  Administration of high-dose chemotherapy in combination with antibodies or target agents would be included in this cohort.
  Interventions: Drug: High intensity therapies

INTERVENTIONS:
Drug: High intensity therapies — * High and intermediate dose Cytarabine
  * Mitoxantrone - Etoposide - Cytarabine (MEC)
  * fludarabine - cytarabine - idarubicin - G-CSF (FLAG-IDA)
  * cladribine - high dose cytarabine (2CDA+HDAraC)
  * mitoxantrone - intermediate dose cytarabine (MiDAC)
  * fludarabine - amsacrine - cytarabine (FLAMSA)
  * Mitoxantrone - Intermediate-dose Cytarabine (HAM)
  * 3+7 (cytarabine and daunorubicine or idarubicine)
  Arms: High intensity treatment
Drug: Low intensity therapies — * Venetoclax+hypomethylating agent (decitabine, azacitidine)
  * Venetoclax+low dose cytarabine
  * Gilteritinib alone or in combination with low dose hypomethylating agent or low dose cytarabine
  * 2CDA 5mg/sqm + low dose cytarabine
  * Glasdegib+low dose cytarabine
  * Ivosidenib alone or in combination with low dose hypomethylating agent or low dose cytarabine
  * Single agent Gemtuzumab or Gemtuzumab in combination with alone or in combination with low dose hypomethylating agent or low dose cytarabine
  Arms: Low intensity treatment

SUMMARY:
This is a multicenter, randomized, open-label, pragmatic low intervention clinical trial comparing high intensity reinduction chemotherapy with low intensity therapies in 1st or 2nd relapse Acute Myeloid Leukemia. The study is funded by European Commission (HORIZON-MISS-2022-CANCER-01-03, Project ID 101104421)

DETAILED DESCRIPTION:
Thanks to recent advantages and results that demonstrate that low-intensity rescues may be quantitatively comparable to chemotherapy, novel personalized therapies are being slowly integrated into the treatment options of R/R AML. These new strategies, for the high interpatient variability, for the different cross-country reimbursement, for the school of thinking of treatment physicians, will wait decades to be proficiently compared with standard chemotherapy in the R/R setting, especially because most of the novel drugs are being pushed by the companies in the front-line (a setting that still has a large room for improvements). In IMPACT-AML RPCT, low-intensity therapies will be compared with high intensity chemotherapy rescue following a pragmatic, clinical-oriented approach. The study is funded by European Commission (HORIZON-MISS-2022-CANCER-01-03, Project ID 101104421)

ELIGIBILITY:
Inclusion Criteria:

* Non-Acute promyelocytic leukemia (APL) AML defined according World Health Organization (WHO) 2022 (or International Consensus Classification (ICC) 2022) criteria
* 1st or 2nd relapse or refractory according to European leukemia Network (ELN) 2022
* Patient is clinically candidate to both low intensity therapy and high dose chemotherapy in the opinion of the physician
* Both low intensity therapy and high dose chemotherapy to which patient is candidate are available and can be provided as per local practice
* No specific treatment protocol can be rationally considered better suited to patient needs.This specifically include, but is not limited to:

  i) the availability of a drug that is already demonstrated superior to comparator arm and can be considered the only standard of care ii) specific contraindications related to fitness or any medical conditions that deem to avoid one of the two arms of this randomization iii) patient willingness to avoid one of the two arm of this randomization iv) lack of social support that make unfeasible one of the two arm of this randomization
* Male or Female, aged>18 years
* Eastern Cooperative Oncology Group (ECOG) performance status <4
* A female participant is eligible to participate if she is not pregnant and not breastfeeding. If Women of childbearing potential (WOCBP), negative serum pregnancy test within 14 days of starting treatment must be obtained. WOCBP must adopt highly effective birth control methods, according to guideline "Recommendation related to contraception and pregnancy testing in clinical trials". Male patient and his female partner who is of childbearing potential must use 2 methods of birth control (a condom as a barrier method of contraception and one of the highly effective birth control methods, according to guideline "Recommendation related to contraception and pregnancy testing in clinical trials". Use of- and compliance to- birth control methods are required beginning at the screening visit and continuing until 6 months following last treatment with study drug.
* Participant is willing and able to give informed consent for participation in the study

Exclusion Criteria:

* Known contraindication to the study drug that will be selected by the treating physician within the list of high or low intensity treatment, according to most update version of Summary of Product Characteristics (SmPC) (e.g. hypersensitivity, allergy, organ failure precluding treatment)
* Participation in another clinical trial with any investigational agents within 14 days or 5 drug half-lives (whatever comes first) prior to randomization
* Active infections or other clinical conditions that in the opinion of the investigator make the patient ineligible to receive study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 339 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
To determine in R/R AML patients the clinical benefit of low intensity therapy as shown by event-free survival compared to high intensity therapy. | 36 months
  Event-free survival defined as time from randomization to treatment failure, hematologic relapse from CR/CRh/Cri or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
To determine if low intensity therapy improves overall survival | 36 months
  Overall survival, defined as time from randomization to the date of death from any cause.
To determine if low intensity therapy improves the overall response (Complete response (CR)/CR with partial hematologic recovery(CRh)/CR with incomplete hematologic recovery(CRi),morphologic leukemia-free state(MLFS)) | 36 months
  Overall response rate (CR/CRh/CRi, MLFS) as the best assessment of response during the study treatment and the overall study cohort.
To determine if low intensity therapy improves patients-reported quality of life | 36 months
  Change in Hematologic Malignancy-Patient-Reported Outcome (HM-PRO) A-total as defined by the HM-PRO questionnaire between screening and end of treatment assessment.
To evaluate the safety of low intensity therapies as compared to high intensity therapies | 36 months
  Proportion of patients experiencing adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Martinelli, MD, Prof, Study Chair — University of Bologna
Locations (36):
- Czechia (5):
  - University Hospital Brno, Brno
  - University Hospital Hradec Králové, Hradec Králové
  - University Hospital Olomouc, Olomouc
  - University Hospital in Ostrava, Ostrava
  - University Hospital in Pilsen, Pilsen
- Germany (6):
  - Uniklinik RWTH Aachen, Aachen
  - University Hospital Greifswald, Greifswald
  - Krankenhaus St. Elisabeth und St. Barbara Halle (Saale) GmbH, Halle
  - University Hospital Halle, Halle
  - University Hospital of Rostock, Rostock
  - Heinrich-Braun-Klinikum gGmbH, Zwickau
- Italy (21):
  - Policlinico Sant'Orsola, Bologna, BO
  - IRCCS Ospedale Policlinico San Martino, Genova, GE
  - Ospedali Riuniti Villa Sofia - Cervello, Palermo, PA
  - Ospedale S.Spirito - ASL Pescara, Pescara, PE
  - Ospedale Santa Maria della Misericordia, Perugia, PG
  - Ospedale Santa Maria delle Croci, Ravenna, RA
  - Policlinico Tor Vergata, Roma, RM
  - Policlinico Umberto I, Roma, RM
  - AOU Città della Salute e della Scienza di Torino, Torino, TO
  - A. O. Ordine Mauriziano, Torino, TO
  - ASST degli Spedali Civili, Brescia
  - ASST Valle Olonda, Busto Arsizio
  - Istituto Oncologico Veneto IRCCS, Castelfranco Veneto
  - AOU Careggi, Florence
  - IRST Istituto Romagnolo per lo Studio dei Tumori Dino Amadori, Meldola
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliera di Rilievo Nazionale Antonio Cardarelli, Napoli
  - Azienda Ospedale-Università Padova, Padua
  - Ospedale Infermi, Rimini
  - Ospedale San Bortolo, Vicenza
- The Hospital of Lithuanian University of Health Sciences Kauno Klinikos, Kaunas, Lithuania
- Hospital de Santa Maria, Lisbon, Portugal
- Fundeni Clinical Institute, Bucharest, Romania
- Instituto de Investigación Sanitaria La Fe, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No